CLINICAL TRIAL: NCT04457011
Title: The Efficacy and Safety Evaluation of Susu Xiao'er Zhike Granules in the Treatment of the Cough Caused by the Common Cold(Wind Cold Cough Syndromes) in Children: a Randomized, Double-blind, Dose Exploration,Multi-center Phase II Clinical Trial
Brief Title: Efficacy and Safety of Susu Zhike Granules for Treating Acute Cough Due to Common Cold With Cold-cough Syndrome in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-SSXEZKKL-Ⅱ
Record Dates: First submitted 2020-06-23; First posted 2020-07-07 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Cough
Keywords: Susu zhike granules
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose group (Experimental): High dose Susu Xiao'er Zhike Granules, 1 bag, bid
  Interventions: Drug: High dose Susu Xiao'er Zhike Granules 1 bag
- Middle dose group (Experimental): Middle dose Susu Xiao'er Zhike Granules, 1 bag, bid
  Interventions: Drug: Middle dose Susu Xiao'er Zhike Granules 1 bag
- Extremely-low dose group (Placebo Comparator): Extremely-low dose Susu Xiao'er Zhike Granules, 1 bag, bid
  Interventions: Drug: Extremely-low dose Susu Xiao'er Zhike Granules 1 bag

INTERVENTIONS:
Drug: High dose Susu Xiao'er Zhike Granules 1 bag — High dose Susu Xiao'er Zhike Granules 1 bag(9g granule per bag,contains 20.25 g crude herbs), twice a day (7-9a.m. and 5-7p.m.) for five days
  Arms: High dose group
Drug: Middle dose Susu Xiao'er Zhike Granules 1 bag — Middle dose Susu Xiao'er Zhike Granules 1 bag(9g granule per bag,contains 10.12 g crude herbs), twice a day (7-9a.m. and 5-7p.m.) for five days
  Arms: Middle dose group
Drug: Extremely-low dose Susu Xiao'er Zhike Granules 1 bag — Extremely-low dose Susu Xiao'er Zhike Granules 1 bag(9g granule per bag,contains 1.01 g crude herbs), twice a day (7-9a.m. and 5-7p.m.) for five days
  Arms: Extremely-low dose group

SUMMARY:
This protocol is designed with the aim of exploring the efficacy of Susu on shortening duration and reducing severity of cough, and observe the safety used in children.

DETAILED DESCRIPTION:
Susu used to be a clinical experienced Chinese herb formula for treating acute cough caused by common cold. The ingredients includes Hua Ju Hong, Qiao Rui Su, Zi Su Ye, Jie Geng, Gan Cao,which relieving cold and cough, resolving phlegm in traditional Chinese medicine theory. This prescription was used for a long time in clinical for treatingacute cough caused by common cold as an herb formula. To standardize the quality and make it easier to take, we reproduced it into a patent medicine and design this trial for evaluating it.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as common cold standard, and VAS score of daytime or night-time cough >= 40mm;
* Diagnosed as wind cold cough syndrome;
* Aged 6-14 ( < 14) years;
* The course of cough is <= 48 hours;
* The maximum temperature is <= 38 degree C within 24 hours before visit;
* The informed consent process complies with the requirement,and the legal representative and the child (>= 8 years old) sign the informed consent form.

Exclusion Criteria:

* Accompanied by sore throat, obvious fever;
* The white blood cell count(WBC), absolute value of neutrophils(NEU) and c-reactive protein(CRP) all exceeded 1.2 times of the upper limit of the reference value, and the researchers considered bacterial infection;
* With complication, such as otitis media, sinusitis, acute bronchitis, pneumonia;
* Acute bronchitis, pneumonia have been cured less than 8 weeks;
* With a medical history of seasonal or perennial allergic rhinitis, chronic sinusitis, chronic otitis media, bronchial asthma, chronic cough or recurrent respiratory tract infection;
* Patients with severe malnutrition;
* Patients with other serious systemic diseases of the cardiovascular, brain, liver, kidney and hematopoietic systems, any anatomical or respiratory abnormalities or mental disorders;
* Allergic to the experimental drugs;
* Received antihistamines or any cough medicine, oral or inhaled steroid preparation before enrollment;
* The investigator considers it inappropriate to participate in this clinical trial.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2020-09-19 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Time to Resolution of cough/ resolution rate | The median time of resolution of cough during Day 2-Day 6 and resolution rate of the last 24 hours.
  Clinical cure is assessed based on visual analogue scale(VAS) score of cough severity, and defined as both VAS scores of day-time and night-time cough reduce to 17mm or less, and last for 24 hours. Day-time refers to 6AM-10PM, night-time refers to 10PM-6AM. The cough VAS is a 100mm line segment, its length represents cough severity (both cough frequent and tense should be considered). 0mm=no cough, 100mm=worst cough, seriously impacting life quality such as playing, going to school, sleeping.18 Day-time and night-time VAS are assessed independently on baseline (Day1) and Day 2-Day 6 to assess the severity of last 24 hours. Children will be trained to use this assessment tool after randomized, and will recorded it by themselves via dairy with the assistance of their parents.

SECONDARY OUTCOMES:
Time to relief of cough | The median time of relief of cough during Day 2-Day 6.
  Day-time and night-time visual analogue scale(VAS) are assessed independently on baseline (Day1) and Day 2-Day 6 to assess the severity of last 24 hours.
Area Under the cough VAS- Time Curve | Baseline(Day1),Day 2-Day 6 post-treatment
  Day-time and night-time visual analogue scale(VAS) are assessed independently on baseline (Day1) and Day 2-Day 6 to assess the severity of last 24 hours.
Parent-proxy Children's Acute Cough-specific QoL Questionnaire(PAC-QoL) scale score | Baseline(Day1),the last 24 hours post-treatment
  PAC-QoL is a 16-iterm parent-proxy questionnaire to reflect the frequency of particular feelings and concerns or worries of parents, developed by team of Sophie Anderson James in Australia. 7 points Lkiert-type scale (very consistent, consistent, some consistent, general, some non-consistent, non-consistent, and very inconsistent, scoring 1-7, respectively) is used to assess the quality of life of past 24 hours. Lower scores shows greater frequency, concerns, or worries, with higher scores therefore reflecting better quality of life.
Overall improvement of cough | The last 24 hours post-treatment
  It is assessed by parents, with the question of "How is your child's cough severity changed after treatment?"(compared with 6 days ago). The response includes much better, better, no difference, worse, much worse. It will be record on Day 6.
Disappearance rate of Traditional Chinese Medicine(TCM) symptom | Baseline(Day1),the last 24 hours post-treatment
  TCM syndrome includes feverish, cough,intolerance of cold, headache, body ache, nasal congestion, sneezing, runny nose, pharyngeal itching.
Curative effect of Traditional Chinese Medicine(TCM) syndrome | Baseline(Day1),the last 24 hours post-treatment
  We will assess the cure rate of symptoms respectively and the total efficacy of traditional Chinese syndrome on Day 6 via the TCM syndrome scale. Cure is defined as the score of the independent symptom decreased to 0. Efficacy means the change from baseline of total score>50%.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Xiamen Hospital of Traditional Chinese Medicine, Xiamen, Fujian
  - Hubei Provincial Hospital of TCM, Wuhan, Hubei
  - The First Hospital of Hunan University of Traditional Chinese Medicine, Changsha, Hunan
  - Shanghai Hospital of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Affiliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - The First Teaching Hospital of Tianjin University of TCM, Tianjin, Tianjin Municipality
  - Yunnan Provincial Hospital of TCM, Kunming, Yunnan